CLINICAL TRIAL: NCT00280917
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of the Safety and Efficacy of Daily CF101 Administered Orally, When Added to Weekly Methotrexate, in Patients With Active Rheumatoid Arthritis
Brief Title: Oral CF101 and Methotrexate Treatment in Rheumatoid Arthritis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Can-Fite BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CF101-202RA
Record Dates: First submitted 2006-01-23; First posted 2006-01-24 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; RA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — CF101

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

INTERVENTIONS:
Drug: CF101

SUMMARY:
This trial will test the hypothesis that the addition of CF101, a novel anti-inflammatory agent, will improve the clinical condition of patients with rheumatoid arthritis who still have active joint inflammation despite taking methotrexate for at least 6 months.

DETAILED DESCRIPTION:
This will be a multi-center, randomized, double-blind, parallel-group, placebo-controlled, dose-finding study in which patients with active RA despite receiving methotrexate for at least 6 months (at unchanged doses for >=2 months) will be randomized to the addition of either CF101 0.1 mg, CF101 1 mg, CF101 4 mg, or placebo given orally q12h for 12 weeks. Screening examinations will occur within 1 month prior to dosing. Washout of other disease-modifying antirheumatic drugs (DMARDs) (with the exception of hydroxychloroquine), including biological agents, will occur prior to dosing; if washout is necessary, patients must re-qualify for inclusion following the washout. Doses of nonsteroidal anti-inflammatory drugs (NSAIDS) and corticosteroids must be stable for >=1 month prior to dosing and remain so during protocol participation. Disease activity will be assessed using swollen and tender joint counts, duration of morning stiffness, physician and patient global assessments (by visual analog scale, VAS), patient reported pain (by VAS), a Health Assessment Questionnaire (HAQ) Disability Index (DI), Westergren erythrocyte sedimentation rate (ESR, Screening, Weeks 0 and12), and C-reactive protein (CRP) levels. Assessments will take place at Screening, Baseline (Week 0), and at Weeks 2, 4, 8, 12, and 14.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 18-75 years
* Meet the criteria of the American Rheumatism Association for RA (Arnett FC et al. Arthritis Rheum 1988;31:315-324, Appendix 1)
* Not bed- or wheelchair-bound
* Active RA, as indicated by the presence of (a) >=6 swollen joints (28 joint count); AND (b) >=6 tender joints (28 joint count); AND at least one of the following: (c) Westergren ESR of >=28 mm/hour; OR (d) CRP level above the upper limit of normal for the central reference laboratory; OR (e) morning stiffness for >=45 minutes
* Treatment with weekly oral or parenteral methotrexate for >=6 months prior to baseline
* Methotrexate route of administration has been unchanged for >=2 months prior to baseline
* Dose of methotrexate has been stable at 15-25 mg/week for >=2 months, and is expected to remain stable throughout the study; the stable dose of methotrexate may alternatively be 10-12.5 mg/week if documented toxicity has precluded a higher dose
* If taking hydroxychloroquine, administration duration has been >=3 months and dose has been stable for >=2 months prior to baseline
* If taking a nonsteroidal anti-inflammatory agent (NSAID), dose has been stable for at least 1 month prior to baseline, and will remain unchanged during protocol participation
* If taking an oral corticosteroid, dose is <=10 mg/day prednisone or equivalent, has been stable for at least 1 month prior to the washout period, and will remain stable through the washout and entire treatment and follow-up period
* Absence of clinically significant findings, such as interstitial pneumonitis or active pulmonary infection, on chest X-ray taken within 6 months prior to screening

Exclusion Criteria:

* Receipt of any of the following for at least a 1 month washout period prior to dosing: sulfasalazine, oral or injectable gold, azathioprine, minocycline, penicillamine, anakinra
* Receipt of etanercept for at least a 6 week period prior to dosing
* Receipt of cyclosporine, infliximab or adalimumab for at least a 2 month period prior to dosing
* Receipt of leflunomide for at least a 2 month period prior to screening, unless patient has undergone cholestyramine washout at least 1 month prior to dosing
* Receipt of cyclophosphamide for at least a 6 month period prior to dosing
* Receipt of rituximab at any previous time
* Receipt of CF101 in a previous trial
* Use of oral corticosteroids >10 mg of prednisone, or equivalent, per day
* Change in NSAID dose level for 1 month prior to dosing
* Change in oral corticosteroid dose level during the 1 month prior to, or during, the washout period
* Change in hydroxychloroquine dose level during the 2 months prior to, or during, the washout period
* Receipt of parenteral or intra-articular corticosteroids during the 1 month prior to, or during, the washout period
* Presence or history of uncontrolled asthma
* Presence or history of uncontrolled arterial hypertension or symptomatic hypotension
* Significant cardiac arrhythmia or conduction block, congestive heart failure, or any other evidence of clinically significant heart disease; other clinically significant findings on screening electrocardiogram (ECG)
* Hemoglobin level <9.0 gm/L
* Platelet count <125,000/mm3
* White blood cell count <3000/mm3
* Serum creatinine level outside the laboratory's normal limits
* Liver aminotransferase levels greater than 1.2 times the laboratory's upper limit of normal
* Known or suspected immunodeficiency or human immunodeficiency virus positivity
* Pregnancy, lactation, or inadequate contraception as judged by the Investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2006-06; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Silverman, MD, Study Director — BioStrategics Consulting Ltd
Locations (27):
- United States (5):
  - Can-Fite Investigational Site, Peoria, Arizona
  - Can-Fite Investigational Site, Albany, New York
  - Can-Fite Invesitigational Site, Cleveland, Ohio
  - Can-Fite Investigational Site, Perrysburg, Ohio
  - Can-Fite Investigational Site, Sugar Land, Texas
- Bulgaria (3):
  - Can-Fite Investigational Site, Plovdiv
  - Can-Fite Investigational Site, Sofia
  - Can-Fite Investigational Site, Stara Zagora
- Israel (7):
  - Can-Fite Investigational Sites, Afula
  - Can-Fite Investigational Site, Ashkelon
  - Can-Fite Investigational Site, Beer Yaakov
  - Can-Fite Investigational Site, Haifa
  - Can-Fite Investigational Site, Jerusalem
  - Can-Fite Investigational Site, Kfar Saba
  - Can-Fite Investigational Site, Tel Litwinsky
- Poland (4):
  - Can-Fite Investigational Site, Bialystok
  - Can-Fite Investigational Site, Lublin
  - Can-Fite Investigational Site, Sopot
  - Can-Fite Investigational Site, Szczecin
- Romania (4):
  - Can-Fite Investigational Site, Brasov
  - Can-Fite Investigational Site, Bucharest
  - Can-Fite Investigational Site, Cluj-Napoca
  - Can-Fite Investigational Site, Iași
- Serbia (3):
  - Can-Fite Investigational Site, Belgrade
  - Can-Fite Investigational Site, Niška Banja
  - Can-Fite Investigational Site, Zemun
- Can-Fite Investigational Site, Kiev, Ukraine

REFERENCES:
- [Background] Szabo C, Scott GS, Virag L, Egnaczyk G, Salzman AL, Shanley TP, Hasko G. Suppression of macrophage inflammatory protein (MIP)-1alpha production and collagen-induced arthritis by adenosine receptor agonists. Br J Pharmacol. 1998 Sep;125(2):379-87. doi: 10.1038/sj.bjp.0702040. PMID 9786512
- [Background] Baharav E, Bar-Yehuda S, Madi L, Silberman D, Rath-Wolfson L, Halpren M, Ochaion A, Weinberger A, Fishman P. Antiinflammatory effect of A3 adenosine receptor agonists in murine autoimmune arthritis models. J Rheumatol. 2005 Mar;32(3):469-76. PMID 15742438

RESULTS

PARTICIPANT FLOW:
Groups:
- CF101 0.1mg: CF101 0.1 mg q12 hours orally
- CF101 1mg: CF101 1mg q12 hours orally
- CF101 4mg: CF101 4mg q12 hours orally
- Placebo: Matching placebo q12 hours orally
Period: Overall Study
Arm/Group | CF101 0.1mg | CF101 1mg | CF101 4mg | Placebo
Started | 65 | 63 | 63 | 63
Completed | 63 | 57 | 57 | 61
Not Completed | 2 | 6 | 6 | 2
Not completed — Adverse Event | 1 | 1 | 4 | 1
Not completed — Change Therapy | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 1
Not completed — Noncompliance | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- CF101 0.1mg: CF101 0.1 mg q12 hours for 12 weeks
- CF101 1mg: CF101 1 mg q12 hours for 12 weeks
- CF101 4mg: CF101 4 mg q12 hours for 12 weeks
- Placebo: Matching Placebo q12 hours for 12 weeks
- Total: Total of all reporting groups
Arm/Group | CF101 0.1mg | CF101 1mg | CF101 4mg | Placebo | Total
Number analyzed (Participants) | 65 | 63 | 63 | 63 | 254
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (12.02) | 54.3 (9.98) | 54.4 (10.07) | 53 (10.86) | 54.1 (10.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 46 | 52 | 52 | 199
  Male | 16 | 17 | 11 | 11 | 55

OUTCOME MEASURES:

1. Primary Outcome: ACR Efficacy Criteria
Description: ACR 20 response (20% improvnent in RA based on swollen and tender joint counts, physician and patient global assessments of disease activity, a patient pain score) at endpoint (Week 12), with all-cause dropouts considered as nonresponders (nonresponder imputation) in the Intent-To-Treat (ITT) population
Time Frame: 12 weeks
Measure: Number; unit: participants
Groups:
- CF101 0.1 mg: CF101 0.1 mg q12 hours for 12 weeks
- CF101 1 mg: CF101 1 mg q12 hours for 12 weeks
- CF101 4 mg: CF101 4 mg q12 hours for 12 weeks
Arm/Group | CF101 0.1 mg | CF101 1 mg | CF101 4 mg | Placebo
Number analyzed (Participants) | 63 | 57 | 57 | 61
participants | 63 | 57 | 57 | 61

2. Secondary Outcome: ACR Criteria Components
Description: ACR 20 response at all visits in the evaluable population and ACR 50 and ACR 70 responses at all visits in the ITT and evaluable populations using both nonresponder imputation and Last Observation Carried Forward (LOCF) analyses; change and percent change from baseline at each visit in the ITT and evaluable populations, analyzed using LOCF, in ACR response components [tender joint count, swollen joint count, patient assessment of pain by VAS, patient global assessment of disease activity by VAS, physician global assessment of disease activity by VAS, HAQ DI, CRP (by central laboratory, using an standard-sensitivity assay capable of detecting changes below the upper limit of normal) and ESR], Disease Activity Score (DAS28), and duration of morning stiffness.
Time Frame: 12 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Safety
Description: Vital signs and weight, physical examinations, adverse event (AE) reporting, clinical laboratory testing, including liver function, renal function, complete blood count and clinical chemistries, urinalysis, and hematologic testing and 12-lead resting ECGs
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- CF101 0.1mg: CF101 0.1 mg given orally q12h for 12 weeks
- CF101 1mg: CF101 1 mg given orally q12h for 12 weeks
- CF101 4mg: CF101 4 mg given orally q12h for 12 weeks
- Placebo: Matching placebo
Arm/Group | CF101 0.1mg | CF101 1mg | CF101 4mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/63 | 2/57 | 2/57 | 0/61
Other Adverse Events (participants affected / at risk) | 0/63 | 0/57 | 0/57 | 0/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CF101 0.1mg (N=63) | CF101 1mg (N=57) | CF101 4mg (N=57) | Placebo (N=61)
PNEUMONIA VIRALIS (Infections and infestations) | 0 | 1 | 0 | 0 — PNEUMONIA VIRAL
hepatitis acute (Infections and infestations) | 0 | 0 | 1 | 0 — Hepatitis B
COPD EXACERBATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 — CHRONIC OBSTRUCTIVE PULMONARY DISEASE
Visual Disturbance (Eye disorders) | 1 | 0 | 0 | 0 — Visual Disturbance
Non small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 — Non small cell lung cancer recurrent
Supposition of Chronic Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 — Bronchitis Chronic

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No